CLINICAL TRIAL: NCT05224128
Title: A Phase I/II, Randomized, Double-Blind Intervention Trial for Evaluating the Safety and Efficacy of Imatinib in Subjects With Advance Fibrosis
Brief Title: Effect of Imatinib in Advance Liver Fibrosis Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Institute for Gastroenterology and Liver Diseases (RIGLD) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1112
Record Dates: First submitted 2022-01-08; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imatinib Drug (Experimental): Standard medication of liver fibrosis + Imatinib 200 mg 1 time a day.
  Interventions: Drug: Imatinib 200mg
- Placebo (Placebo Comparator): Standard medication of liver fibrosis + placebo as a control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imatinib 200mg — Imatinib have to be taken 200mg/day orally for 24 weeks in a seated position with a meal or a large (at least 250 mL) glass of water
  Other Names: Trade name Gleevec or other name STI-571
  Arms: Imatinib Drug
Drug: Placebo — Capsules (similar appearance with imatinib) without active substance have to be taken orally for 24 weeks in a seated position with a meal or a large (at least 250 mL) glass of water
  Arms: Placebo

SUMMARY:
When a recurrent, long-term injury and inflammation of the liver causes an excessive accumulation of damaged tissue, a dangerous condition called liver fibrosis develops. Most chronic liver diseases eventually lead to fibrosis. Activated hepatic stellate cells (aHSC) play an important role in the development of hepatic fibrosis. Inhibiting the proliferation of stellate cells and preventing their differentiation and activation is an ideal strategy for ameliorating hepatic fibrosis. Hence imatinib have been prescribed as a promising drug to limit the progression of liver fibrosis as a clinical inhibitor of tyrosine kinase which can affect the two main pathways leading to hepatic stellate cells activation.

DETAILED DESCRIPTION:
Liver fibrosis can be categorized as a serious health problem worldwide. It is widely recognized that activated hepatic stellate cells (HSC) play a pivotal role in pathological development of liver fibrosis. The activated hepatic stellate cells (aHSCs) are main producers of ECM, which play a significant role in scarring process of the liver derived from variety of etiologies, such as hepatitis B or C virus infection, chronic alcohol abuse, non-alcoholic steatohepatitis, cholestasis, and autoimmune hepatitis. Due to lack of effective treatments, chronic liver diseases and liver fibrosis can eventually progress to liver cirrhosis and even liver cancer. Inhibition of the stellate cell proliferation, differentiation and prevention of its activation is appealing as an ideal strategy for ameliorating hepatic fibrosis. A platelet-derived growth factor (PDGF) is the most potent proliferating stimulus for HSC. Imatinib mesylate (Gleevec), a clinically used PDGF receptor (PDGFR) tyrosine kinase inhibitor could be a promising molecular targeted approach to limit the liver fibrosis development. IL-6/STAT3 is one the pivotal signaling pathways for the activation of HSCs. Herein in our previous study we found that Imatinib upregulates miR-124 and interferes simultaneously with STAT3-HLF-IL-6 pathway. However, due to effective role of imatinib in blocking two important liver fibrosis related pathways, pharmacokinetics of imatinib in patients with liver fibrosis have never been assessed. This study is a phase I/II, double blind labeled, randomized, double arms clinical trial. Consequently, this phase I/II trial was initiated to evaluate the safety and efficacy of imatinib in patients with advanced liver fibrosis. 20 patients with clinical and/or pathologic diagnosis of liver fibrosis grade 3-4 will be registered at Taleghani hospital (Tehran). 10 patients will receive standard medication and imatinib for 24 weeks at the dose of 200mg/day orally. Another 10 patients will be treated with standard medication of liver fibrosis and placebo of imatinib drug as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between18-75 years old with a clinically confirmed diagnosis of Fibrosis with grade 3-4 by Metavir score.
* BMI >25
* Negative alcohol screen
* Able to understand and willing to voluntarily sign an informed consent form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

* Known cardiovascular disease.
* Requiring any of the following medications during the duration of the study:History of cirrhosis based on imaging or clinical criteria and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding.
* History of hepatocellular carcinoma (HCC)
* History of malignancy within the past 5 years or ongoing malignancy other than basal cell carcinoma, or resected noninvasive cutaneous squamous carcinoma at the time of Screening visit.
* Active, serious infections that requires parenteral antibiotic or antifungal therapy within 30 days prior to Screening visit.
* Females who are pregnant or breastfeeding.
* Current or anticipated treatment with radiation therapy, cytotoxic chemotherapeutic agents and immunomodulating agents (such as systemic corticosteroids, interleukins, interferons).
* Use of any experimental medications within the last 6 months of Screening Visit.
* Familial dyslipidemia Weight loss of >5% within 6 months prior to Screening, based on subject's reporting Currently or participated in a weight loss program within the last 6 months.
* Any history of bariatric surgery Diabetes mellitus Type I.
* Daily alcohol intake >20 ml (2 units)/day for women and 30 ml (3 units)/day for men (on average), as per Alcohol Use Disorders Identification Test (AUDIT) questionnaire at Screening and plan to consume the same alcohol amount referenced above during the trial.
* Use of any immunosuppressive medication, anti-inflammatory monoclonal antibody treatment, or chronic systemic corticosteroids >10 mg prednisone-equivalent concurrently or within 1 year prior to Screening.
* Uncontrolled or clinically unstable thyroid disease, in the judgment of the Principal Investigator.
* History or presence of hepatitis B or C or human immunodeficiency virus (HIV) Uncontrolled arterial hypertension.
* Any severe, acute, or chronic medical or psychiatric condition that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or in compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the subject inappropriate for entry into this study.
* Subjects who have previously received imatinib or who have history of hypersensitivity, allergy, intolerance or contraindication to imatinib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-02-02 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of liver fibrosis score changes from baseline to 6 months | 6 months
  by the FibroScan system

SECONDARY OUTCOMES:
Alanine aminotransferase serum levels changes in baseline, 3 months and 6months | every 3 months for 6 months
  Serology testing
Aspartate aminotransferase serum levels changes in baseline, 3 months and 6months | every 3 months for 6 months
  Serology testing
Albumin levels changes in baseline, 3 months and 6months | every 3 months for 6 months
  Serology testing
Bilirubin levels changes in baseline, 3 months and 6months | every 3 months for 6 months
  Serology testing
Detecting changes of Tumor necrosis factor (TNF)-alpha from baseline to 6 months | 6 months
  Serology testing of the serum inflammation markers
Detecting changes of Interleukin-6 from baseline to 6 months | 6 months
  Serology testing of the serum inflammation markers
Blood sugar changes in baseline, 3 months and 6months | every 3 months for 6 months
  Blood test
Fasting insulin changes in baseline, 3 months and 6months | every 3 months for 6 months
  Blood test
Complete blood count changes in baseline, 3 months and 6months | every 3 months for 6 months
  Blood test
International normalized ratio (INR) changes in baseline, 3 months and 6months | every 3 months for 6 months
  Blood test
Prothrombin time (PT) changes in baseline, 3 months and 6months | every 3 months for 6 months
  Blood test

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Gastroenterology & Liver Diseases, Tehran, Iran